CLINICAL TRIAL: NCT02407275
Title: ETUDE DU MICROBIOTE DES RHINOSINUSITES CHRONIQUES DIFFICILES A TRAITER PAR METAGENOMIQUE ET CULTUROMIQUE
Brief Title: Rhinosinusites Chroniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Hospitalo-Universitaire Méditerranée Infection (Other)
Collaborators: University Hospital, Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IHU Méditerranée Infections
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Sinusitis; Chronic Disease; Refractory
MeSH Terms: conditions — Sinusitis; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- biological sample (Other): Genomic & culturomic analyses
  Interventions: Other: Biological sample

INTERVENTIONS:
Other: Biological sample

SUMMARY:
To analyse and describe sinus microbiota, during hard to treat (or refractory) rhinosinusitis, using culturomic and metagenomic methods (i.e. to culture on many different medium of culture to grow hard to cultivate bacteria + to sequence and analyse all DNA contained in samples).

Samples are middle meatus swabs or pus aspiration, done during usually patient following.

ELIGIBILITY:
Inclusion Criteria:

* >18 year old
* chronic refractory rhinosinusitis
* to require middle meatus swab or other sinus sample
* absence of opposition

Exclusion Criteria:

* <18 year old
* pregnant women
* breastfeeding
* under trusteeship
* under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Sinusian microbiota description | 6 months
  species, number and type of isolated microbes

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Edouard Fournier, Professor, Study Chair — IHU Méditerranée Infection
Locations (1):
- Service ORL et de Chirurgie Cervico - Faciale/ AP-HM, Marseille, France